CLINICAL TRIAL: NCT07303920
Title: Wear Experience With Daily Disposable Contact Lenses for Astigmatism Over a Long-Wear Day
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Jennifer Fogt, Assistant Professor, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20252462
Record Dates: First submitted 2025-12-23; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Contact Lens Wear (Other): All participants will be fit with the study contact lenses for astigmatism
  Interventions: Device: Daily disposable contact lenses for astigmatism

INTERVENTIONS:
Device: Daily disposable contact lenses for astigmatism — All participants will be fit with the study lenses
  Other Names: Dailies Total1 for Astigmatism

SUMMARY:
The purpose of this study to assess the wear experience of people who have astigmatism when wearing a daily disposable contact lens for astigmatism over long days of wear.

ELIGIBILITY:
Inclusion Criteria:

* Current soft toric contact lens wearer with long hours of wear
* Willing to follow the contact lens wearing schedule required by the study
* Vision 20/25 or better with current soft toric contact lenses
* Self-report completion of a comprehensive eye examination in the past two years

Exclusion Criteria:

* Have a history of corneal ocular surgery
* Have current ocular inflammation or infection as assessed by the study investigator who will complete the study
* Are past rigid contact lens wearers
* Have a history of being diagnosed with dry eye or ocular allergies
* Have known systemic health conditions that are thought to alter tear film physiology
* Have a history of viral eye disease
* Have a history of ocular surgery
* Have a history of severe ocular trauma
* Have a history of corneal dystrophies or degenerations
* Have active ocular infection or inflammation
* Are currently using isotretinoin-derivatives or ocular medications
* Are pregnant or breast feeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Comfort | Measured over 16 hours of wear
  Proportion of participants with positive Visual Analog Scale (VAS, >50 on a 0-100 scale)

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University College of Optometry, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No